CLINICAL TRIAL: NCT02741245
Title: A Phase III, Randomized, Active Comparator-controlled, Clinical Trial to Study the Efficacy and Safety of MK-0653H in Japanese Patients With Hypercholesterolemia.
Brief Title: A Study of the Efficacy and Safety of MK-0653H in Japanese Participants With Hypercholesterolemia (MK-0653H-832)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653H-832; 163336 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ezetimibe 10 mg (Active Comparator): 1 Ezetimibe 10 mg tablet and 2 Rosuvastatin placebo capsules once daily for 12 weeks
  Interventions: Drug: Ezetimibe 10 mg; Drug: Placebo for Rosuvastatin
- Rosuvastatin 2.5 mg (Active Comparator): 1 Rosuvastatin 2.5 mg capsule, 1 Rosuvastatin placebo capsule and 1 Ezetimibe placebo tablet once daily for 12 weeks.
  Interventions: Drug: Rosuvastatin 2.5 mg; Drug: Placebo for Ezetimibe; Drug: Placebo for Rosuvastatin
- Rosuvastatin 5.0 mg (Active Comparator): 2 Rosuvastatin 2.5 mg capsules and Ezetimibe placebo tablet once daily for 12 weeks.
  Interventions: Drug: Rosuvastatin 2.5 mg; Drug: Placebo for Ezetimibe
- Ezetimibe 10 mg+ Rosuvastatin 2.5 mg (Experimental): 1 Ezetimbie 10 mg tablet, 1 Rosuvastatin 2.5 mg capsule and 1 Rosuvastatin placebo capsule once daily for 12 weeks.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Rosuvastatin 2.5 mg; Drug: Placebo for Rosuvastatin
- Ezetimibe 10 mg+ Rosuvastatin 5.0 mg (Experimental): 1 Ezetimbie 10 mg tablet and 2 Rosuvastatin 2.5 mg capsules once daily for 12 weeks.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Rosuvastatin 2.5 mg

INTERVENTIONS:
Drug: Ezetimibe 10 mg
  Arms: Ezetimibe 10 mg; Ezetimibe 10 mg+ Rosuvastatin 2.5 mg; Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Drug: Rosuvastatin 2.5 mg
  Arms: Ezetimibe 10 mg+ Rosuvastatin 2.5 mg; Ezetimibe 10 mg+ Rosuvastatin 5.0 mg; Rosuvastatin 2.5 mg; Rosuvastatin 5.0 mg
Drug: Placebo for Ezetimibe
  Arms: Rosuvastatin 2.5 mg; Rosuvastatin 5.0 mg
Drug: Placebo for Rosuvastatin
  Arms: Ezetimibe 10 mg; Ezetimibe 10 mg+ Rosuvastatin 2.5 mg; Rosuvastatin 2.5 mg

SUMMARY:
This study will evaluate the efficacy and safety and tolerability of 2 dose levels of MK-0653H in Japanese participants. The primary hypotheses are that the administration of MK-0653H is safe and tolerable and that MK-0653H is superior to single entity of Ezetimibe and Rosuvastatin in percent reduction from baseline in low-density lipoprotein-cholesterol (LDL-C) after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Japanese
* Outpatient with hypercholesterolemia
* Female participant who is of reproductive potential has to agree to remain abstinent or use (or partner use) two acceptable methods of birth control from date of signed informed consent to the 14 days after the last dose of study drug
* Will maintain a stable diet that is consistent with the Japan Atherosclerosis Society Guideline 2012 (JAS 2012) for prevention of atherosclerotic cardiovascular diseases for the duration of the study

Exclusion Criteria:

* Uncontrolled hypertension (treated or untreated)
* Uncontrolled type 1 or type 2 diabetes mellitus
* History of coronary artery disease (CAD), CAD-equivalent disease
* Familial hypercholesterolemia or has undergone LDL apheresis
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Has had a gastrointestinal tract bypass, or other significant intestinal malabsorption
* History of cancer within the past 5 years (except for successfully treated dermatological basal cell or squamous cell carcinoma or in situ cervical cancer)
* Human Immunodeficiency Virus (HIV) positive
* History of drug/ alcohol abuse within the past 5 years or psychiatric illness not adequately controlled and stable on pharmacotherapy
* Consumes more than 25 g of alcohol per day
* Currently following an excessive weight reduction diet
* Currently engages in a vigorous exercise regimen (e.g.; marathon training, body building training etc.) or intends to start training during the study
* Hypersensitivity or intolerance to Ezetimibe or Rosuvastatin
* Myopathy or rhabdomyolysis with Ezetimibe or any statin
* Pregnant or lactating
* Taking any other investigational drugs and/or has taken any investigational drugs within 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teramoto T, Yokote K, Nishida C, Oshima N, Takase T. A phase III clinical trial to study the efficacy and safety of ezetimibe plus rosuvastatin combination therapy in Japanese patients with hypercholesterolemia - A randomized, double-blind comparative study. J Clin Therapeut Med. 2017;33(11):881-896.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Started | 35 | 72 | 71 | 71 | 72
Completed | 35 | 71 | 71 | 67 | 70
Not Completed | 0 | 1 | 0 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg | Total
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72 | 321
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (8.9) | 55.7 (10.6) | 58.9 (9.0) | 56.0 (10.3) | 58.2 (10.6) | 57.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 36 | 40 | 37 | 37 | 166
  Male | 19 | 36 | 31 | 34 | 35 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 35 | 72 | 71 | 71 | 72 | 321
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 35 | 72 | 71 | 71 | 72 | 321
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Low-density Lipoprotein-cholesterol (LDL-C)
Description: Participants had LDL-C levels assessed at baseline and after 12 weeks of study drug administration. The change from baseline was calculated. Results were reported as a M-estimate.
Time Frame: Baseline and Week 12
Population: All randomized participants who received at least 1 dose of study drug, had baseline or post-baseline data and had baseline data for those analyses that required baseline data.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage Change | -18.7 [-21.9 to -15.5] | -39.8 [-42.0 to -37.5] | -47.2 [-49.4 to -44.9] | -54.6 [-56.9 to -52.3] | -60.5 [-62.8 to -58.2]
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Ezetimibe 10 mg+ Rosuvastatin 2.5 mg; Test type: Other; p < 0.001, Shapiro-Wilk test; Robust regression model with terms for treatment, risk category and baseline, after imputing missing values by a multiple imputation approach; Difference in M-estimates = -35.9, 95% CI 2-sided [-39.9 to -32.0]
Statistical Analysis 2: Comparison: Rosuvastatin 2.5 mg vs Ezetimibe 10 mg+ Rosuvastatin 2.5 mg; Test type: Other — Robust regression model with terms for treatment, risk category and baseline, after imputing missing values by a multiple imputation approach; p < 0.001, Shapiro-Wilk test; Difference in M-estimates = -14.8, 95% CI 2-sided [-18.0 to -11.6]
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Ezetimibe 10 mg+ Rosuvastatin 5.0 mg; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.001, Shapiro-Wilk test; Difference in M-estimates = -41.8, 95% CI 2-sided [-45.8 to -37.9]
Statistical Analysis 4: Comparison: Rosuvastatin 5.0 mg vs Ezetimibe 10 mg+ Rosuvastatin 5.0 mg; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.001, Shapiro-Wilk test; Differecne in M-estimates = -13.3, 95% CI 2-sided [-16.6 to -10.1]

2. Primary Outcome: Percentage of Participants Who Experience at Least 1 Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized
Time Frame: up to 14 weeks
Population: All randomized participants who received at least 1 dose of doubleblind study treatment and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 31.4 | 34.7 | 42.3 | 40.8 | 37.5

3. Primary Outcome: Percentage of Participants Who Had Study Drug Discontinued Due to Adverse Event
Description: An AE was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. The percentage of participants that had study drug discontinued due to an AE was summarized.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of participants | 0.0 | 0.0 | 0.0 | 2.8 | 1.4

4. Primary Outcome: Percentage of Participants Who Experience 1 or More Gastrointestinal-related AEs
Description: Gastrointestinal-related AEs included all preferred terms within system organ class of Gastrointestinal Disorders except Chapped Lips and Toothache.
Time Frame: up to 14 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 6.9 | 4.2 | 8.5 | 2.8

5. Primary Outcome: Percentage of Participants Who Experience 1 or More Gallbladder-related AEs
Description: Gallbladder-related AEs included Bile Duct Obstruction, Bile Duct Stone, Bile Duct Stenosis, Biliary Colic, Cholangitis, Cholecystectomy, Cholecystitis, Cholelithiasis, Gallbladder Disorder, Gallbladder Perforation, Hepatic Pain, and Hydrocholecystis.
Time Frame: up to 14 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants Who Experience 1 or More Allergic Reaction or Rash AEs
Description: Allergic Reaction or Rash AEs included Allergy to Arthropod Sting, Anaphylactoid Reaction, Anaphylactic Reaction, Anaphylatic Shock, Anaphylactoid Shock, Angioedema, Conjunctivitis Allergic, Contrast Media Reaction, Dermatitis, Dermatitis Allergic, Dermatitis Atopic, Dermatitis Bullous, Dermatitis Contact, Dermatitis Psoriasiform, Drug Hypersensitivity, Eczema, Eosinophila, Erythema, Eye Allergy, Face Oedema, Hypersensitivity, Mechanical Urticaria, Palmar Erythema, Periorbital Oedema, Photodermatosis, Photosensitivity Allergic reaction, Photosensitivity Reaction, Pigmentation Disorder, Pruritus, Pruritus Generalised, Rash, Rash Erythematous, Rash Follicular, Rash Generalised, Rash Maculo-Papular, Rash Papulosquamous, Rash Pruritic, Rash Pustular, Rash Vesicular, Rhinitis, Rhinitis Allergic, Rosacea, Skin Exfoliation, Skin Disorder, Skin Hyperpigmentation, Skin Lesion, Skin Mass, Skin Ulcer, Subcutaneous Nodule, Swelling Face, Systemic Lupus Erythematosus Rash, Urticaria.
Time Frame: up to 14 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 1.4 | 4.2 | 2.8 | 2.8

7. Primary Outcome: Percentage of Participants Who Experience 1 or More Hepatitis-related AEs
Description: Hepatitis-related AEs included Cholestasis, Cytolytic Hepatitis, Hepatic Cyst, Hepatic Failure, Hepatic Lesion, Hepatic Necrosis, Hepatitis, Hepatitis Cholestatic, Hepatitis Fulminant, Hepatitis Infectious, Hepatocellular Injury, Hepatomegaly, Jaundice, Jaundice Cholestatic.
Time Frame: up to 14 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in Alanine Aminotransferase (ALT) ≥3 Times Upper Normal Limit (ULN)
Description: Participants had ALT levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of ALT that were 3 x ULN or greater were recorded. The ALT ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.4 | 0.0

9. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in Aspartate Aminotransferase (AST) ≥3 Times Upper Normal Limit (ULN)
Description: Participants had AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of AST that were 3 x ULN or greater were recorded. The AST ULN was 40 U/L..
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

10. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) ≥3 Times Upper Normal Limit (ULN)
Description: Participants had ALT and AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of ALT and/or AST that were 3 x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.4 | 0.0

11. Primary Outcome: Percentage of Participants Who Experience Elevation in Alanine Aminotransferase (ALT) ≥5 Times Upper Normal Limit (ULN)
Description: Participants had ALT levels assessed throughout the 12 week treatment period. Participants who had an assessments of ALT that was 5x ULN or greater were recorded. The ALT ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

12. Primary Outcome: Percentage of Participants Who Experience Elevation in Aspartate Aminotransferase (AST) ≥5 Times Upper Normal Limit (ULN)
Description: Participants had AST levels assessed throughout the 12 week treatment period. Participants who had an assessments of AST that was 5x ULN or greater were recorded. The AST ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

13. Primary Outcome: Percentage of Participants Who Experience Elevation in Alanine Aminotransferase (ALT) ≥10 Times Upper Normal Limit (ULN)
Description: Participants had ALT levels assessed throughout the 12 week treatment period. Participants who had an assessments of ALT that was 10x ULN or greater were recorded. The ALT ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

14. Primary Outcome: Percentage of Participants Who Experience Elevation in Aspartate Aminotransferase (AST) ≥10 Times Upper Normal Limit (ULN)
Description: Participants had AST levels assessed throughout the 12 week treatment period. Participants who had an assessments of AST that was 10x ULN or greater were recorded. The AST ULN was 40 U/L.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

15. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) ≥10 Times Upper Normal Limit (ULN)
Description: Participants had ALT and AST levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of ALT and/or AST that were 10x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

16. Primary Outcome: Percentage of Participants With Potential Hy's Law Condition
Description: Percentage of Participants with Potential Hy's Law Condition (defined as serum ALT or serum AST elevations >3xULN, with serum alkalinephosphatase <2xULN and total bilirubin (TBL) ≥2xULN) was summarized. The ALT and AST ULNs were 40 U/L. The ULN for alkaline phosphatase was 359 IU/L and the ULN for total bilirubin was 1.2 mg/dL.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

17. Primary Outcome: Percentage of Participants Who Experience Elevations in Creatine Kinase (CK) ≥10 Times ULN
Description: Participants had creatine phosphokinase (CK) levels assessed throughout the 12 week treatment period. Participants who had any CK level that was ≥10 x ULN were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

18. Primary Outcome: Percentage of Participants Who Experience Elevations in Creatine Kinase (CK) ≥10 Times ULN With Muscle Symptoms
Description: Participants had CK levels assessed throughout the 52 week treatment period. Participants who had any CK level that was ≥10 x ULN and had associated muscle symptoms present within +/- 7 days were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

19. Primary Outcome: Percentage of Participants Who Experience Elevations in Creatine Kinase (CK) ≥10 Times ULN and Drug-Related Muscle Symptoms
Description: Participants had CK levels assessed throughout the 52 week treatment period. Participants who had any CK level that was ≥10 x ULN and had associated muscle symptoms present within +/- 7 days that were reported as at least possibly-related to study drug were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
Number analyzed (Participants) | 35 | 72 | 71 | 71 | 72
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: up to 2 weeks post last dose of study drug (up to 14 weeks total)
Description: All participants that received at least 1 dose of study drug.
Arm/Group | Ezetimibe 10 mg | Rosuvastatin 2.5 mg | Rosuvastatin 5.0 mg | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/72 | 0/71 | 0/71 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/72 | 1/71 | 0/71 | 0/72
Other Adverse Events (participants affected / at risk) | 6/35 | 8/72 | 11/71 | 6/71 | 7/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg (N=35) | Rosuvastatin 2.5 mg (N=72) | Rosuvastatin 5.0 mg (N=71) | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg (N=71) | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg (N=72)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg (N=35) | Rosuvastatin 2.5 mg (N=72) | Rosuvastatin 5.0 mg (N=71) | Ezetimibe 10 mg+ Rosuvastatin 2.5 mg (N=71) | Ezetimibe 10 mg+ Rosuvastatin 5.0 mg (N=72)
Nasopharyngitis (Infections and infestations) | 6 (6) | 8 (9) | 11 (12) | 6 (6) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT02741245/Prot_SAP_000.pdf